CLINICAL TRIAL: NCT05640232
Title: A National, Multicenter, Randomized, Double-blind, Double-dummy, Phase III, Crossover Study to Assess the Efficacy and Safety of CDE100 in the Treatment of Menstrual Cramp Pain Associated With Primary Dysmenorrhea.
Brief Title: Efficacy and Safety of CDE100 in the Treatment of Menstrual Cramp Pain Associated With Primary Dysmenorrhea
Acronym: ASTRAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMS0522 - ASTRAL
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, Double-dummy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): CDE100 The patient must take 1 pill of CDE100 association and placebo of Buscopan® Composto association, if pain, until three times a day.
  Interventions: Drug: CDE100 association
- Control (Active Comparator): Buscopan® Composto association.
  The patient must take 1 pill of Buscopan® Composto association and placebo of CDE100 association, if pain, until three times a day.
  Interventions: Drug: Buscopan® Composto association

INTERVENTIONS:
Drug: CDE100 association — Experimental drug.
  Arms: Experimental
Drug: Buscopan® Composto association — Active comparator.
  Arms: Control

SUMMARY:
The purpose of this study if to evaluate the efficacy and safety of CDE100 in the Treatment of Menstrual Cramp Pain Associated With Primary Dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent to participate in the study prior to admission to the study;
* Female patients aged between 16 and 35 years old, inclusive;
* History of regular menstrual cycles, occuring between every 21 to 35 days;
* Clinical history compatible with the diagnosis of primary dysmenorrhea;
* Self-reported history of ≥ 4 painful cycles, with moderate or severe menstrual cramps, in the six (06) months prior to selection for the study.

Exclusion Criteria:

* Diagnosis of secondary dysmenorrhea;
* History of non-response to treatment with non-steroidal anti-inflammatory drugs (NSAIDs) to relieve menstrual cramps;
* Onset of primary dysmenorrhea after starting to use oral contraceptives;
* Use of oral contraceptives for < 3 months prior to study selection;
* Use of an intrauterine device (IUD), hormonal implants or contraceptive injections in the last six (06) months;
* Previous diagnosis or physical examination findings and/or clinical and/or surgical history that may indicate the presence of endometriosis, pelvic inflammatory disease, adenomyosis, mullerian duct malformation, uterine fibroma, cystic ovary and/or pelvic varicocele;
* History of recurrent pelvic and/or lower abdominal pain outside the menstrual period;
* Presence of known allergy or hypersensitivity to the components of the drugs used during the clinical trial;
* History of hypersensitivity reactions, such as asthma attacks or other types of allergic reactions, to acetylsalicylic acid or other NSAIDs;
* History or diagnosis of peptic/hemorrhagic ulcer;
* History of gastrointestinal bleeding or perforation related to the use of NSAIDs;
* Presence of compromised bone marrow function or diseases of the hematopoietic system;
* Diagnosis of acute intermittent hepatic porphyria;
* Diagnosis of congenital deficiency of glucose-6-phosphate dehydrogenase (G6PD);
* Diagnosis of untreated angle-closure glaucoma;
* Presence of mechanical stenosis in the gastrointestinal tract;
* Diagnosis of megacolon and/or paralytic or obstructive ileus;
* Diagnosis of myasthenia gravis;
* Treatment with psychoactive drugs (such as, for example, antidepressants, antipsychotics, etc.) in the 30 days prior to selection for the study;
* Participants with a history of alcohol or illicit drug use disorder in the last two (02) years;
* Participants with a current medical history of cancer and/or cancer treatment in the last five (05) years;
* Presence of any serious illness, at the discretion of the investigator;
* Any finding of clinical observation (clinical/physical evaluation) or laboratory condition that is interpreted by the investigating physician as a risk to the participation of the research participant in the clinical trial or presence of uncontrolled chronic disease(s);
* Participants who are pregnant, nursing or planning to become pregnant;
* Disagreement with the use of a known effective barrier contraceptive method, unless using a stable oral contraceptive for three months or more (which must be maintained throughout the study), or surgically sterile or who expressly declare themselves exempt from risk of pregnancy for not exercising sexual practices or exercising them in a non-reproductive manner;
* Participation in a clinical research protocol in the last 12 months (CNS Resolution 251, of August 7, 1997, item III, subitem J), unless the investigator judges that there may be a direct benefit to it;
* Presence of any condition that, at the discretion of the investigator, makes the patient unfit to participate in the study.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Women with moderate to severe pain associated with primary dysmenorrhea.
Enrollment: 238 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Sum of Total Pain Relief (TOTPAR) over 0-4 hours post-dose. | 4 hours post-dose.
  Pain relief will be evaluated considering the Sum of Total Pain Relief (TOTPAR) over 0-4 hours post-dose. Pain relief will be evaluate using a Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief).

SECONDARY OUTCOMES:
Sum of Total Pain Relief (TOTPAR) over 0-8 hours post-dose. | 8 hours post-dose.
  Pain relief will be evaluated considering the Sum of Total Pain Relief (TOTPAR) over 0-8 hours post-dose. Pain relief will be evaluate using a Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief).
Sum of Pain Intensity Difference (SPID) over 4 hours post-dose. | 4 hours post-dose.
  Sum of Pain Intensity Difference (SPID) over 4 hours post-dose. The pain intensity will be assessed using a Categorical 4-point scale (0 = no pain, 1 = mild pain, 2 = moderate pain, 3 = severe pain).
Sum of Pain Intensity Difference (SPID) over 8 hours post-dose. | 8 hours post-dose.
  Sum of Pain Intensity Difference (SPID) over 8 hours post-dose. The pain intensity will be assessed using a Categorical 4-point scale (0 = no pain, 1 = mild pain, 2 = moderate pain, 3 = severe pain).
Time to first intake of rescue medication. | Up to 8 hours post-dose.
  Time between the first dose intake and the administration of a rescue medication.
Patients who used rescue medication. | Up to 8 hours post-dose.
  Number of participants who used rescue medication after the first drug intake.
Doses of rescue medication used. | Up to 8 hours post-dose.
  Number of rescue medication doses used in the first day of treatment.
Number of additional drug intake. | 3 days.
  Number of additional drug intake during the study period.
Patients' Global Impression of Change (PGIC). | 8 hours.
  Patients' Global Impression of Change (PGIC) will be assessed after 8 hours post-dose or immediately before the intake of rescue medication.
Evaluate the safety of CDE100 association in the treatment of primary dysmenorrhea. | Up to 175 days.
  The safety will be evaluated considering the incidence of adverse events (AEs) reported during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- EMS, Hortolândia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No